CLINICAL TRIAL: NCT04295122
Title: Comparing the Effectiveness of Phacoemulsification + ECP Laser and Phacoemulsification Alone for the Treatment of Open Angle Glaucoma in Patients With Cataract - a Randomised Controlled Trial
Brief Title: Comparing the Effectiveness of Phacoemulsification + ECP Laser and Phacoemulsification Alone for Glaucoma Patients
Acronym: CONCEPT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 263262
Record Dates: First submitted 2020-02-25; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Glaucoma Open-Angle Primary; Cataract
Keywords: Glaucoma; Cataract; ECP laser
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract; Glaucoma | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phacoemulsification + ECP laser (Active Comparator): Cataract surgery will be performed using standard anesthesia and phacoemulsification techniques. A clear corneal incision should be used for instrumentation. The choice of viscoelastics to maintain the anterior chamber is left to the surgeon's discretion. The viscoelastic will be washed-out of the capsular bag after IOL insertion. Further cohesive viscoelastic material will be injected through the main wound between the anterior capsule and iris, until the iris is close to or touching the cornea. A curved ECP probe will be inserted through the corneal incision wound/wounds and 360° of the anterior section of the ciliary processes will be treated. The power setting will be varied according to tissue response (starting power of 250 mW with continuous setting). 'Pops' should be avoided (but recorded) but no indentation used during treatment.
  Intracameral cefuroxime and dexamethasone will be injected into the anterior chamber and sutures used to close the incisions as required.
  Interventions: Device: Phacoemulsification+ Endoscopic cyclophotocoagulation (ECP) laser
- Phacoemulsification alone (Active Comparator): Cataract surgery will be performed using standard anesthesia and phacoemulsification techniques. A clear corneal incision should be used for instrumentation. The choice of viscoelastics to maintain the anterior chamber is left to the surgeon's discretion. For this study, monofocal IOLs are required.
  Interventions: Device: Phacoemulsification+ Endoscopic cyclophotocoagulation (ECP) laser

INTERVENTIONS:
Device: Phacoemulsification+ Endoscopic cyclophotocoagulation (ECP) laser — A clear corneal incision should be used for instrumentation. The choice of viscoelastics to maintain the anterior chamber is left to the surgeon's discretion.
  Phacoemulsification energy used during the cataract surgery will be recorded. If the patient has been randomised to ECP laser, the viscoelastic will be washed-out of the capsular bag. Further cohesive viscoelastic material will be injected through the main wound between the anterior capsule and iris, until the iris is close to or touching the cornea. A curved ECP probe will be inserted through the corneal incision wound/wounds and 360° of the anterior section of the ciliary processes will be treated. The power setting will be varied according to tissue response (starting power of 250 mW with continuous setting). 'Pops' should be avoided (but recorded) but no indentation used during treatment. Final power used and duration of surgery will be recorded.

SUMMARY:
Laser endoscopic cyclophotocoagulation (ECP) has been in use for the treatment of glaucoma for over 20 years and is usually used in conjunction with cataract surgery. In the US it is one of the most commonly performed cataract 'plus' surgeries. The take-up of ECP laser has been much lower in the UK and Europe. This is partly due to the lack of robust clinical evidence from randomised controlled trials to justify its use in routine practice. More recently the advent of minimally invasive glaucoma surgery techniques (MIGS) has increased the options available for cataract 'plus' surgery. Without any randomised controlled trial data for the use of ECP laser in this context the increasingly popular use of MIGS devices, such as iStent (the current market leader) may further marginalise the use of ECP laser for cataract 'plus' surgery in patients with Primary Open Angle Glaucoma (POAG) and visually significant cataract.

To further evaluate the use of ECP laser for the treatment of glaucoma in patients with glaucoma and cataract, investigators plan to conduct a randomised controlled trial comparing cataract surgery alone versus cataract surgery plus ECP laser surgery. Investigators will compare the efficacy of these interventions for the treatment of glaucoma based on clinical outcomes and also undertake a cost-benefit analysis, taking into account the cost of surgery, any reduction in clinical time allocation for procedures, the frequency of intra- and post-operative complications, and any reduction in the need for topical glaucoma treatments post-surgery, as well as the frequency with which further glaucoma filtering surgery is needed for patients in each group.

Investigators anticipate that a total number of 160 patients (80 in each arm) will be adequate to detect whether there is any difference in efficacy between cataract surgery + ECP versus cataract surgery alone. Recruitment is expected to take around 9-12 months. Participants will undergo treatment wash-out (28 days minimum) of any eye drops they use for their glaucoma prior to data collection at baseline (before surgery) and prior to data collection at one-year and at two-years post-surgery. Results will be reviewed during an interim analysis at 6 months once 50 patients have reached that time point.

DETAILED DESCRIPTION:
The study compares one off surgical interventions that are in routine clinical use and therefore there are no major ethical issues. All participants will be eligible for cataract surgery. Participants will be randomly allocated to one or other of the treatment arms. Explicit written consent for randomisation will be obtained and recorded on the consent form. The available evidence does not indicate that there are substantially greater risks of intra- and post-operative complications associated with combined ECP plus cataract surgery compared with cataract surgery alone.

Participants may be asked to attend an additional visit for the baseline pre-operative data collection. The tests undertaken at this visit would therefore be additional non-routine procedures. If the baseline data collection is undertaken at an additional, rather than a routine visit, then travel expenses to will be paid for the extra non-routine visit.

At the some visits additional tests will be performed that would not normally be routinely undertaken with glaucoma patients at those visits. All of the tests that will be done for the study are routinely performed in ophthalmology out-patient clinics, but the non-routine tests may not be routinely performed with glaucoma patients or may not be routinely performed at all visits.

Participants will be asked to stop using their eye drops for glaucoma at least 28 days before the pre-operative baseline measurements are taken and again at least 28 days before the 1 year and 2 years post-operative measurements are taken (if they continue to need eye drops after surgery). This will not cause participants any harm and will not have a clinical impact on their glaucoma or their vision. Including a treatment washout period is common practice in glaucoma research. If it is not clinically safe for a patient to stop taking the eye drops they use to treat their glaucoma or ocular hypertension for 4 weeks, or if they are not willing to stop using their eye drops for 4 weeks, then they will be excluded from the study. To minimise risk only patients with mild to moderate glaucoma will be included. Those with advanced disease will be excluded. The treatment washout will not cause any delay to the surgery as the usual waiting time for surgery is 1-2 months.

To be on the safe side some participants may be asked to come in two weeks after stopping taking their eye drops so the investigators can do a safety check of the pressure in their eyes. Most patients who take part in the study will not need this. If investigator do ask a participant to come in for a safety check this will be an extra appointment that they would not normally be asked to come to if the participant were not taking part in the study, so the travel expenses will be paid. It will be a brief appointment (10-15 minutes) to check the intraocular pressure by Goldmann applanation tonometry. This is the standard test for intraocular pressure that is performed at all routine glaucoma clinic visits. Participants may potentially need to come in for three IOP safety check visits if a washout is required before the 1 year and 2 years follow-up visits because treatment by eye drops is continued after surgery.

Participants will be asked to come to the all of the appointments that they would be asked to attend if they were not taking part and will receive the same post-operative clinical care that they would receive if not taking part.

Benefits

There are no benefits to participants. However, the study aims to help us to understand more about how best to treat glaucoma and as relatives of people with glaucoma have a higher than normal risk of developing glaucoma, the study could in the future be of benefit to participants' relatives.

2. Trial design and statistics

2.1 Trial Design The study will be a single blinded prospective randomised two armed surgical trial to compare the effectiveness and cost effectiveness of phacoemulsification combined with ECP laser versus phacoemulsification alone for the treatment of early or moderate open angle glaucoma (OAG) in patients with visually significant cataract eligible for phacoemulsification (cataract surgery). Treatment allocation will be masked for participants. As the study team includes the surgeons who perform the surgical procedures the investigators will not be masked as to which treatment the patient receives.

Settings

This study will be conducted in the Ophthalmology Department at St Thomas' Hospital (Guy's and St Thomas' NHS Foundation Trust). Other sites in the UK will be invited to participate if the recruitment rate is below expectation.

Trail duration Patients will be recruited for 9-12 months up to a maximum of 160 patients (with up to 80 allocated to each arm). Patients' participation will last for up to 2 years and 6 months consisting of a maximum of 60 days from screening/enrolment to the commencement of treatment washout, a maximum of 60 days treatment washout, a maximum of 60 days from the baseline measurements to surgery, and then 2 years post-operative follow-up. The total study duration with therefore be up to 3 years and 6 months (up to 12 months recruitment plus up to 2 years and 6 months for the last participant to complete the study).

2.3 Outcome Measures Primary outcome - change in post-washout IOP of at least 2.7 mmHg at 12 and 24 months from baseline. The IOP will be measured using Goldmann applanation tonometer at each visit.

Secondary outcomes:

1. The % of patients with reduction of mean diurnal IOP of ≥ 20% from baseline at 24 months following medication washout. (Note: throughout this protocol, the term "diurnal IOP" is synonymous with "washed out diurnal IOP".)
2. Change in number of glaucoma medication used at 24 months from baseline.
3. Cost effectiveness. This will be assessed by collecting the flowing parameters:

   1. Time needed for surgery.
   2. Time for personnel (process mapping).
   3. Cost of laser. Other Measures
   4. Clinic visits (patient questionnaire).
   5. GP visits (patient questionnaire).
   6. Pharmacy visits (patient questionnaire).
   7. Medications (patient questionnaire).
   8. Further glaucoma surgery (patient questionnaire). If yes, which one? How many?
   9. Complication related to the initial surgery (operation note and CRF review).
4. Intra- and Post - operative complication rates:

   Safety outcomes include:
   * Loss of > 2 lines of BCVA.
   * Slit lamp and fundus examination findings.
   * The incidence of complications and adverse events.

   2.4 Trial statistics and analysis

   Power Calculation and Sample Size Estimate

   A sample size of 58 in each group will have 90% power to detect a difference in means of 2.7 (the difference between a Group 1 mean, µ₁, of 4.5 and a Group 2 mean, µ₂, of 1.8) assuming that the Group 1 standard deviation, σ₁, is 5.13 and the Group 2 standard deviation, σ₂, is 3.61 (ratio of Group 2 to Group 1 standard deviation is 0.704) using a two group Satterthwaite t-test with a 0.05 two-sided significance level.

   Allowing for up to 20% loss to follow-up, 80 patients in each arm will be required for this study, with a total number of 160 patients.

   Statistical Analysis Baseline characteristics of the groups will be summarised with means and standard deviations for continuous data (normally distributed) or medians and inter quartile ranges (non-normal) and numbers with percentages for categorical variables. Outcomes will be reported in a similar fashion again by treatment group.

   Treatment differences will be estimated with 95% confidence intervals analysed. Investigators will analyse on an ITT basis. Missing data will be evaluated and summarised by reason. Should data be missing investigators will report the reasons for this and assess whether or not it appears related to treatment status. Where participants are withdrawn or choose to withdraw prior to randomisation they will not be included in the final analysis.

   Cost Effectiveness Analysis (UK Model)

   The cost effectiveness analysis will look at the current care pathway and outline how ECP laser will affect the time taken to do a procedure by understanding the current standard of care for a Glaucoma patient post operatively and costs associated at each stage. Formulating a quantitative care pathway model will effectively assess how ECP laser could allow for cost benefits within the NHS. The secondary focus of this RCT will be look at current standards and compare how time and resources can be effectively reduced by implementing ECP laser. A budget impact model can be created once the RCT complete and data for cost benefit which will be used for payer groups. The cost benefit will look at the following below:
   * Time reductions - If using ECP as the new standard of care (instead of drainage surgery), time reductions operatively will allow for more surgical procedures to be performed in theatres, which will benefit NHS Trusts.
   * Change in number of glaucoma therapeutic drugs - Cost savings can be naturally made if the surgical procedure is sustainable over a period of 2 years.

   Criteria for discontinuation/early withdrawal of participants from the study

   Failure to meet eligibility criteria prior to randomisation

   Enrolled patients may be withdrawn from the study during the pre-baseline treatment washout, after the baseline data collection and after cataract surgery if they are ineligible to continue in the study according to the following criteria:
   * During pre-baseline treatment washout (before randomization): If treatment washout is stopped at an IOP safety check visit during the pre-baseline treatment washout the participant will be withdrawn except in cases where the fellow eye is eligible for inclusion, in which case they may remain in the study.
   * At baseline (before randomization): If the IOP in the study eye is outside the specified range (18 mmHg & 40 mmHg inclusive) at baseline the participant would be withdrawn except in cases where the fellow eye is eligible for inclusion, in which case they may remain in the study.
   * After cataract surgery (before randomization): If cataract surgery is complicated or a physical pupil dilatation device is used during surgery (i.e. the procedure is not an uncomplicated cataract surgery and IOL implantation) then the participant will not be randomized and will be withdrawn except in cases where the fellow eye is eligible for inclusion, in which case they may remain in the study.

   Because enrolled participants may not meet the above criteria for continuing in the study up to randomization, a significant percentage of participants are expected to exit the study prior to qualifying for surgery and randomization.

   Where participants are withdrawn prior to randomization because they do not meet the above protocol defined criteria for remaining in the study:
   * No further data will be collected from them for the study and they will not be included in the final analysis.
   * Safety events that occur prior to withdrawal will be recorded and any patient with a safety event will not be exited from the study until the event is resolved or stable.
   * These patients will not be required to undergo further study related examinations.

   Where a participant's treatment washout is stopped on an IOP safety check visit during their treatment washout before the 1 or 2 year follow up visits (i.e. post randomisation) then they will not be withdrawn but the post-washout data will be treated as missing data.

   Other grounds for early withdrawal from the study

   Patients' participation in the study is entirely voluntary and each participant has the right to withdraw from the study at any time.

   In addition, the investigator may discontinue a participant from the study at any time if the investigator considers it necessary for any reason, including:
   * Ineligibility (either arising during the study or retrospectively, having been overlooked at screening).
   * Significant protocol deviation.
   * An adverse event which results in the participant being unable to continue to comply with study procedures.
   * Disease progression which results in the participant being unable to continue to comply with study procedures.
   * If in the opinion of the investigator, the study procedures threaten the health or well-being of the patient.
   * Consent withdrawn or loss of capacity.
   * Lost to follow up.
   * Inability to continue
   * At patient's request

   Notification of a patient's early termination should be made immediately to the Sponsor and documented on the appropriate CRF.

   Where participants are withdrawn or choose to withdraw prior to randomisation any data collected will not be included in the final analysis.

   Patients who are withdrawn or choose to withdraw from the study will not be replaced (the sample size includes an estimate of the likely number of participants who may be withdrawn due to failure to meet the criteria for staying in the study up to randomisation).

   Where participants are withdrawn or choose to withdraw for any reason:
   * The reason for withdrawal will be recorded.
   * Data collected up to that point will be retained but no further data will be collected.
   * Decisions about their surgery and future clinical care after withdrawal will be based on usual clinical practice. They will not be treated according to the study protocol.
   * Enrolled patients with an adverse event will be followed-up until resolution or stabilisation of the event. If the participant is withdrawn due to an adverse event the investigator will arrange for follow-up visits or telephone calls until the adverse event has resolved or stabilised.

   Participants lost to follow-up

   Patients who cannot be successfully contacted after several attempts will be considered lost to follow-up. Contact attempts will consist of the following:
   * Three (3) documented phone calls and/or e-mails, followed by
   * One (1) certified letter. Patients who are lost to follow-up will not be replaced; however, patients may be recovered if contact is re-initiated at any time prior to the patient's 2 years' follow-up visit.

   Study procedures and data to be collected at each visit

   Appendix A summarizes the procedures to be conducted at each study visit.

   Baseline

   Baseline assessments will be undertaken after 28-60 days treatment washout (i.e. at a minimum 29 days from the commencement of treatment washout) and no more than 60 days before surgery. The baseline visit may be an additional (i.e. non-routine) visit. All tests and procedures performed at this visit are therefore additional procedures not routine care. The procedures to be conducted at the baseline visit and the data to be recorded are detailed below:
   * Eligibility review including a check of all exclusion criteria to ensure that none apply and baseline IOP criteria.
   * Demographic details (date of birth and age, gender, ethnicity).
   * Medical history/significant diagnoses
   * Details of any ocular or other medications.
   * Ophthalmic examination. The following procedures will be performed and the findings recorded:

     * Refraction/Auto-refraction
     * Snellen Visual Acuity
     * Slit Lamp Biomicroscopy (examination of the eye)
     * Tonometry/IOP measurement (Goldmann applanation tonometry will be used to measure IOP. The IOP measurement will be done after application of topical anesthetic (eye drop) with fluorescein): IOP will be measured at two time-points: 9AM +/- 2 hours and 11AM +/- 2 hours
     * Pachymetry / central corneal thickness
     * Gonioscopy
     * Perimetry (Visual field test) (Humphrey Field Analyzer, HFA II, automated white on white, 24-2 SITA-standard, Carl Zeiss Meditec Inc., Dublin, CA, USA)
     * OCT scan of optic discs and macular
     * Biometry: Anterior chamber depth and axial length
   * Assessment and recording of any postoperative complications or other adverse events.
   * Assessment and recording of any need for supplemental medical therapy or additional glaucoma surgery.

   Day 0/Surgery

   The procedures to be conducted on the day of surgery and the data to be recorded are detailed below:
   * Eligibility review including a check of all exclusion criteria to ensure that none apply.
   * Details of any ocular or other medications.
   * Surgery:

     * The surgery actually performed will be documented.
     * Any other comments/events in relation to the surgery will also be documented.
     * The phacoemulsification energy used during the cataract surgery will be recorded.
     * ECP procedure: The final power used and duration of surgery will be recorded, and 'Pops' recorded.
   * Randomization
   * The reasons for withdrawal will be documented where patients are withdrawn from the study before randomization because they do not meet all the intra-operative eligibility criteria after cataract surgery.
   * Ophthalmic examination. The following procedures will be performed and the findings recorded:

     - Snellen Visual Acuity
     * Slit Lamp Biomicroscopy
     * Tonometry/IOP measurement
   * Assessment and recording of any intra-operative or postoperative complications or other adverse events.
   * Assessment and recording of any need for supplemental medical therapy or additional glaucoma surgery.

   Follow-up assessments The follow up period for the study is two years. Participants will be followed up at clinic visits by members of the research team in a dedicated ophthalmology research area or in the glaucoma clinic. The need for continued follow-up and timely visits will be stressed to the patient throughout the study.

   The schedule for follow up visits will be the same as would be the case for normal clinical care. Data will be collected at 1 day (range 1-3 days), 1 week (range 5-9 days), 1 month (range 3-5 weeks), 3 months (range 10-14 weeks), 6 months (range 21-26 weeks), 1 year (range 337-407 days), and 2 years (range 680-728 days) post-operative.

   Appendix A summarises the procedures to be conducted at each of the scheduled follow up visits. The procedures to be conducted at the post-operative routine follow-up visits and the data to be recorded are detailed below:
   1. Day, 1 week, 1 month, 3 months and 6 months follow-up • Eligibility review including a check of all exclusion criteria to ensure that none apply.

      * Details of any ocular or other medications.
      * Ophthalmic examination (as per usual care). The following procedures will be performed and the findings recorded:

        - Refraction/Auto-refraction

        o Not performed at 1 day follow-up.

        o Routine at 1 week and 1 month follow-up only.

        o Additional non-routine procedure at 3 months and 6 months follow-up.

        - Snellen Visual Acuity (as per usual care).

        - Slit Lamp Biomicroscopy (as per usual care).
        * Tonometry/IOP measurement (as per usual care).
        * Perimetry (Visual field test) at 6 months follow-up only (as per usual care). Not performed at 1 Day, 1 week, 1 month, and 3 months follow-up.
      * Assessment of the success or failure of the surgery (at 6 months follow-up only).
      * Assessment and recording of any postoperative complications or other adverse events.
      * Assessment and recording of any need for supplemental medical therapy or additional glaucoma surgery.

   <!-- -->

   1. year and 2 years follow-up • Eligibility review including a check of all exclusion criteria to ensure that none apply.

      • Medical history/significant diagnoses (at 1 year follow-up only)

      • Details of any ocular or other medications.

      • Ophthalmic examination (as per usual care). The following procedures will be performed and the findings recorded:

      - Snellen Visual Acuity (as per usual care).

      - Slit Lamp Biomicroscopy (as per usual care).

      - Tonometry/IOP measurement: At 1 and 2 years follow-up IOP will be measured at two time-points: 9AM +/- 2 hours and 11AM +/- 2 hours. At both visits the first IOP measurement is as per usual care but the second IOP measurement is a non-routine procedure).

      - Gonioscopy (as per usual care).
      * Perimetry (Visual field test) (as per usual care).
      * OCT scan of optic discs and macular (as per usual care).
      * Refraction/Auto-refraction (non-routine procedure at 1 and 2 years follow-up)
      * Pachymetry / central corneal thickness (non-routine procedure at 1 and 2 years follow-up)
      * Biometry: Anterior chamber depth and axial length (non-routine procedure at 1 and 2 years follow-up).

        • Assessment of the success or failure of the surgery.

        • Assessment and recording of any postoperative complications or other adverse events.
        * Assessment and recording of any need for supplemental medical therapy or additional glaucoma surgery.
        * At the final visit (2 years post-operative) participants may be told whether or not they had the ECP laser procedure as well as cataract surgery.

      8.1 Unscheduled visits and additional procedures Where participants attend any unscheduled appointments the date and reason for the visit will be recorded on a CRF.

      Details of any additional procedures will also be recorded on a CRF (type of procedure, date, reason for procedure being undertaken).

      8.2 Definition of End of Trial The end of the trial is defined as the date of the last follow-up visit for data collection of the last patient participating in the study. At this point the REC will be informed that the study has been completed by way of an end of study notification.

      8.3 Criteria for the early termination of the trial It is not anticipated that there will be any grounds for early termination of the study. All participants will be eligible for phacoemulsification (cataract surgery). Both phacoemulsification and the ECP laser procedures are already routinely performed. The ECP laser procedure would not normally be done together with phacoemulsification, so for those participants allocated to the phacoemulsification plus ECP arm, ECP will be an extra non-routine procedure. However, the available evidence does not indicate that there are substantially greater risks of intra- and post-operative complications associated with combined phacoemulsification plus ECP compared with phacoemulsification alone.

      No study interventions will be undertaken during the follow up period. During follow up the only deviation from normal care is that additional eye tests will be performed at the 12 weeks and 1 and 2 years post-operative follow-up assessments (routine appointments) and any participants still taking eye drops for their glaucoma after the surgery will be asked to stop taking their eye drops (treatment washout) for a minimum of 4 weeks before the 1 and 2 years post-operative follow-up assessments. All of the eye tests that will be performed for the study are routinely used in the Ophthalmology Department.

      8.4 Source Data

      The source documents from which participants' CRF data will be obtained (i.e. the original documents, data, and records) will include:
      * Patients' hospital records (from which medical history and previous and concurrent medication may be summarised into the CRF).
      * Glaucoma clinic notes.
      * Data / printouts from eye tests conducted during the study and earlier. All documents will be stored safely in confidential conditions. On all study-specific documents, other than the signed consent, the participant will be referred to by the study participant number/code, not by name.

   9 Safety Reporting Also see APPENDIX B: Information with regards to Safety Reporting in Non-CTIMP Research.

   9.1 Definitions Adverse Event (AE) An adverse event (AE) is any untoward medical occurrence in a patient (or other clinical investigation participant taking part in a trial of a medical device) which does not necessarily have to have a causal relationship with the device under investigation.

   An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of the device, whether or not considered related to the device.

   Adverse Device Effect (ADE) Adverse device effects (ADEs) are all untoward and unintended responses to the medical device. The phrase 'responses to the medical device' means that a causal relationship between the device under investigation and an AE is at least a reasonable possibility (i.e. the relationship cannot be ruled out).

   All cases judged by either the reporting medically qualified professional or the sponsor as having a reasonable suspected causal relationship to the device qualify as a device effect.

   This also includes any event resulting from insufficiencies or inadequacies in the instruction(s) for use or deployment of the device and includes any event that is a result of a user error.

   Serious Adverse Event (SAE):

   A serious adverse event (SAE) is an adverse event that:
   * Led to death
   * Led to fetal distress, fetal death, congenital abnormality or birth defect. (Note that pregnant women and women with child bearing potential, including if not using contraceptives, are excluded.)
   * Led to serious deterioration in the health of the patient that - resulted in a life-threatening illness or injury, [NOTE: The term 'life-threatening' in the definition of 'serious' refers to an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe.] - resulted in a permanent impairment of a body structure or a body function,

     * required in-patient hospitalisation or the prolongation of existing hospitalisation, or
     * resulted in medical or surgical intervention to prevent permanent impairment to a body structure or a body function.

   Other important medical events that may not result in death, are not life threatening, or do not require hospitalisation, may be considered a serious adverse event when, based upon appropriate medical judgement, the event may jeopardise the patient and may require medical or surgical intervention to prevent one of the outcomes listed above.

   To ensure no confusion or misunderstanding of the difference between the terms 'serious' and 'severe', which are not synonymous, the following note of clarification is provided:

   The term 'severe' is often used to describe the intensity (severity) of a specific event (as in mild, moderate, or severe myocardial infarction). The event itself, however, may be of relatively minor medical significance (such as severe headache). This is not the same as 'serious', which is based on patient/event outcome or action criteria usually associated with events that pose a threat to a participant's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

   Serious Adverse Device Effects (SADE):

   A serious adverse device effect (SADE) is any untoward medical occurrence seen in a patient that can be attributed wholly or partly to the device and which resulted in any of the characteristics of, or led to a characteristic of, a serious adverse event.

   A SADE is also any event that may have led to these consequences if suitable action had not been taken or an intervention had not been made, or if circumstances had been less opportune.

   All cases are judged by either the reporting medically qualified professional or the sponsor.

   Unanticipated Adverse Device Effect (UADE):

   A unanticipated adverse device effect (UADE) is any serious adverse device effect on health or safety or any life-threatening problem or death caused by, or associated with a device, if that effect, problem, or death was not previously identified in nature, severity or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problem associated with a device that related to the rights, safety or welfare of the patient.

   9.2 Reporting of Adverse Events All AE's occurring during the study observed by the investigator or reported by the participant, whether or not attributed to the device under investigation will be recorded on the CRF as specified in the protocol. All ADE's will be recorded in the CRF.

   The following information will be recorded: description, date of onset and end date, severity, assessment of relatedness to device, other suspect drug or device and action taken. Follow-up information should be provided as necessary.

   The relationship of AEs to the device will be assessed by a medically qualified investigator or the sponsor/manufacturer and will be followed up until resolution or the event is considered stable.

   All ADE that result in a participant's withdrawal from the study or are present at the end of the study, should be followed up until a satisfactory resolution occurs.

   Any pregnancy occurring during the clinical study will be recorded. 9.3 Reporting Procedures for All Adverse Events For studies of CE marked devices all SAE/SADE/UADEs need to be reported to the sponsor/legal representative (in this case Guy's and St Thomas' NHS Foundation Trust) and the device manufacturer (BVI) and Guy's and St Thomas' NHS Foundation Trust (GSTT) within one working day of the investigator team becoming aware of them.

   Reports of related and unexpected SAEs should be submitted to ethics within 15 days of the Chief Investigator becoming aware of the event, using the SAE report form for non-CTIMPs published on the NRES website.

   All reporting to GSTT R&D should be by fax (0207 188 8330) giving as much information about the incident as possible, and should be signed by the PI or Co-investigator. The Guy's and St Thomas' NHS Foundation Trust (GSTFT) SADE reporting form should be used for GSTT sponsored studies.

   The GSTT R&D Department will undertake an initial review of the information and ensure it is reviewed by GSTT R&D. Events will be followed up until resolution and any appropriate further information will be sent by the research team in a timely manner.

   Reporting to the MHRA will be done in liaison with the Chief Investigator and the Manufacturer.

   The Manufacturer has a legal obligation to report all events that need to be reported to the Nominated Competent Authority immediately (without any unjustifiable delay) after a link is established between the event and the device, but no more than:
   * 2 days following the awareness of the event for Serious Public Health Threat.
   * 10 days following awareness of the event for Death or unanticipated serious deterioration in health.
   * 30 days following the awareness of the event for all other event meeting the SAE criteria.

   9.4 Annual Reports In addition to the above reporting the Chief Investigator will submit a progress/safety report to the REC and R&D once a year (or on request) throughout the trial.

   9.5 Criteria for the Termination of the Trial The study compares one off surgical interventions that are currently in routine clinical use in the department. It is not anticipated that any situation will arise that requires termination of the trial.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria:

1. Male and female patients, from 40 to 85 years of age, inclusive.
2. Patient is able and willing to attend scheduled follow-up examinations as per routine care for 2 year post-operatively.
3. Patient is able to understand the information sheet and give informed consent.

   Inclusion criteria for the study eye:
4. An operable age-related cataract with BCVA of 6/9 or worse that is eligible for phacoemulsification.
5. A diagnosis of POAG or pigmentary glaucoma treated with hypotensive medications (eye drops for glaucoma).
6. A previously documented unmedicated intraocular pressure of > 21 mmHg (i.e. IOP > 21 mmHg prior to the commencement of glaucoma treatment).
7. An optic nerve appearance characteristic of glaucoma with either:

   1. visual field loss (no worse than -12dB) identified on examination using Humphrey 24-2 SITA standard, or
   2. (in patients where the VF exam is not confirmatory for glaucomatous defect) OCT retinal nerve fibre layer imaging supporting the ophthalmoscopy findings indicating a diagnosis of mild glaucoma. (If OCT findings are not confirmatory of glaucoma and both the visual field and the OCT are normal, the patient should not be enrolled).
8. Shaffer grade ≥2 in all four quadrants on gonioscopy.
9. Absence of peripheral anterior synechiae (PAS), rubeosis or other angle abnormalities that could impair surgical access to the ciliary processes.

Exclusion Criteria:

1. Diagnosis of Primary angle closure glaucoma.
2. Any diabetic retinopathy.
3. Previous history of Central Serous Retinopathy or Cystoid Macular Oedema in either eye.
4. Congenital or developmental glaucoma.
5. Secondary glaucoma (such as neovascular, uveitic, pseudoexfoliative, lens-induced, steroid-induced, trauma induced, or glaucoma associated with increased episcleral venous pressure).
6. Previous trabeculectomy, tube shunts, or any other prior subconjunctival filtration or cycloderstructive surgery.
7. Inability to complete a reliable 24-2 SITA Standard Humphrey visual field on the study eye at screening (fixation losses, false positive errors and false negative errors should not be greater than 33%).
8. Patients with advanced glaucoma or any patient where the risk to the patient of a washout of ocular hypotensive medications (eye drops for glaucoma) is assessed as unacceptable (i.e. where there may be a risk of damage to vision if treatment is stopped for the washout).
9. Best corrected visual acuity worse than 6/36 in the fellow eye (i.e. not the eye undergoing the study intervention).
10. A 24-2 SITA Standard Humphrey visual field mean deviation (MD) of worse than -12dB in the study eye.
11. Previous vitreo-retinal surgery.
12. Previous corneal surgery or clinically significant corneal dystrophy, e.g. Fuch's dystrophy (>12 confluent guttae).
13. Unclear ocular media preventing visualization of the fundus or anterior chamber angle.
14. Degenerative visual disorders such as wet age-related macular degeneration.
15. Clinically significant ocular pathology other than cataract and glaucoma.
16. Clinically significant ocular inflammation or infection within 1 month prior to screening.
17. Presence of extensive iris processes that obscure visualization of the trabecular meshwork.
18. Uncontrolled systemic disease that in the opinion of the investigator would put the patient's health at risk and/or prevent the patient from completing all study visits.
19. Current participation or participation within the past 30 calendar days in another investigational drug or device clinical trial (which includes the fellow eye).
20. Pregnant or nursing women, or women of child bearing age planning pregnancy or not using medically acceptable contraceptives.
21. Unwilling or unable to give informed consent/unwilling to accept randomisation.
22. Unwilling or unable to return for scheduled protocol visits.
23. Any inclusion criteria not met.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-03-15 (Estimated); Primary Completion 2022-03-14 (Estimated); Study Completion 2023-03-14 (Estimated)

PRIMARY OUTCOMES:
Change in post-washout IOP at 24 months | Two years
  Change in post-washout IOP of at least 2.7 mmHg at 24 months from baseline. The IOP will be measured using Goldmann applanation tonometer at each visit.

SECONDARY OUTCOMES:
The percentage of IOP reduction | Two years
  The % of patients with reduction of mean diurnal IOP of ≥ 20% from baseline at 24 months following medication washout.The IOP will be measured using Goldmann applanation tonometer at 9 am and 11 am at baseline, 12 and 24 months follow up visits. Mean diurnal IOP will be calculated using statistics package.
Change in number of glaucoma medication used | Two years
  Change in number of glaucoma medication used at 24 months from baseline.
Cost effectiveness | Two years
  Time reductions - If using ECP as the new standard of care (instead of drainage surgery), time reductions operatively will allow for more surgical procedures to be performed in theatres, which will benefit NHS Trusts.
  Change in number of glaucoma therapeutic drugs - Cost savings can be naturally made if the surgical procedure is sustainable over a period of 2 years. Clinic, GP and pharmacy visits required will be assessed using patient questionnaire.
Intra- and Post-operative complication rates | Two years
  Rate of complications will be recorded and compared between two groups. Safety outcomes include: Loss of > 2 lines of BCVA, slit lamp and fundus examination findings, the incidence of complications and adverse events.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] The Advanced Glaucoma Intervention Study (AGIS): 7. The relationship between control of intraocular pressure and visual field deterioration.The AGIS Investigators. Am J Ophthalmol. 2000 Oct;130(4):429-40. doi: 10.1016/s0002-9394(00)00538-9. PMID 11024415
- [Background] AGIS Investigators. The Advanced Glaucoma Intervention Study (AGIS): 9. Comparison of glaucoma outcomes in black and white patients within treatment groups. Am J Ophthalmol. 2001 Sep;132(3):311-20. doi: 10.1016/s0002-9394(01)01028-5. PMID 11530042
- [Background] Comparison of glaucomatous progression between untreated patients with normal-tension glaucoma and patients with therapeutically reduced intraocular pressures. Collaborative Normal-Tension Glaucoma Study Group. Am J Ophthalmol. 1998 Oct;126(4):487-97. doi: 10.1016/s0002-9394(98)00223-2. PMID 9780093
- [Background] Kass MA, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, Parrish RK 2nd, Wilson MR, Gordon MO. The Ocular Hypertension Treatment Study: a randomized trial determines that topical ocular hypotensive medication delays or prevents the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002 Jun;120(6):701-13; discussion 829-30. doi: 10.1001/archopht.120.6.701. PMID 12049574
- [Background] Konstas AG, Maskaleris G, Gratsonidis S, Sardelli C. Compliance and viewpoint of glaucoma patients in Greece. Eye (Lond). 2000 Oct;14 Pt 5:752-6. doi: 10.1038/eye.2000.197. PMID 11116698
- [Background] Brown MM, Brown GC, Spaeth GL. Improper topical self-administration of ocular medication among patients with glaucoma. Can J Ophthalmol. 1984 Feb;19(1):2-5. PMID 6608974
- [Background] Gedde SJ, Feuer WJ, Shi W, Lim KS, Barton K, Goyal S, Ahmed IIK, Brandt J; Primary Tube Versus Trabeculectomy Study Group. Treatment Outcomes in the Primary Tube Versus Trabeculectomy Study after 1 Year of Follow-up. Ophthalmology. 2018 May;125(5):650-663. doi: 10.1016/j.ophtha.2018.02.003. Epub 2018 Feb 21. PMID 29477688
- [Background] Gedde SJ, Herndon LW, Brandt JD, Budenz DL, Feuer WJ, Schiffman JC. Surgical complications in the Tube Versus Trabeculectomy Study during the first year of follow-up. Am J Ophthalmol. 2007 Jan;143(1):23-31. doi: 10.1016/j.ajo.2006.07.022. Epub 2006 Sep 1. PMID 17054896
- [Background] Katz LJ. A call for innovative operations for glaucoma. Arch Ophthalmol. 2000 Mar;118(3):412-3. doi: 10.1001/archopht.118.3.412. No abstract available. PMID 10721967
- [Background] Shields MB. Cyclodestructive surgery for glaucoma: past, present, and future. Trans Am Ophthalmol Soc. 1985;83:285-303. PMID 3832531
- [Background] Bloom PA, Dharmaraj S. Endoscopic and transscleral cyclophotocoagulation. Br J Ophthalmol. 2006 Jun;90(6):666-8. doi: 10.1136/bjo.2005.082073. PMID 16714260
- [Background] Pastor SA, Singh K, Lee DA, Juzych MS, Lin SC, Netland PA, Nguyen NT. Cyclophotocoagulation: a report by the American Academy of Ophthalmology. Ophthalmology. 2001 Nov;108(11):2130-8. doi: 10.1016/s0161-6420(01)00889-2. PMID 11713091